CLINICAL TRIAL: NCT05382585
Title: A Cohort Study to Identify Newer Therapeutic Targets in Head and Neck Cancers
Brief Title: Newer Therapeutic Targets in Head and Neck Cancers
Status: Recruiting | Type: Observational
Sponsor: Banaras Hindu University (Other)
Responsible Party: Principal Investigator, Manoj Pandey, Professor, Banaras Hindu University
Other Study IDs: NGSHN1
Record Dates: First submitted 2022-05-16; First posted 2022-05-19 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Head Neck Cancer; Oral Cancer
Keywords: Next generation sequencing; predictive biomarker
MeSH Terms: conditions — Head and Neck Neoplasms; Mouth Neoplasms | interventions — High-Throughput Nucleotide Sequencing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Paraffin embedded tissue
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Head neck cancer: Histologically diagnosed cases of head and neck cancer
  Interventions: Other: Next generation Sequencing

INTERVENTIONS:
Other: Next generation Sequencing — Next generation sequencing for 161 genes

SUMMARY:
Based on the recently identified mutations in HNSCCs, the major pathologic pathways implicated in the tumorigenesis of HNSCC include dysregulation of four processes:

1. cellular survival and proliferation (e.g., TP53, EGFR, MET, and PIK3CA);
2. cell-cycle control (e.g., CDKN2A and CCND1);
3. cellular differentiation (e.g., NOTCH1); and
4. Adhesion and invasion signaling (e.g., FAT1).7 TP53, EGFR, PIK3CA, CDKN2A, CCND1, and MET participate in several common signaling pathways.

Alterations of these genes are most frequently seen in alcohol and tobacco-related HNSCC. However their role in prognostication and selection of therapeutics is not known

DETAILED DESCRIPTION:
Sample size:

Patients with squamous cell carcinoma of oral cavity fulfilling the inclusion and exclusion criteria and willing to participate will be included in this study.

Method:

Comprehensive history and physical examination of the patients will be carried out and all the details will be recorded in the preset proforma. All routine investigations as indicated including a biopsy to establish a diagnosis and CT of the head and neck to measure the tumor dimensions and stage the disease before initiation of treatment will be recorded. The paraffin embedded tissue will be studied for expression of various genetic mutations using NGS platform. Brush cytology will be collected in liquid medium for HPV typing using PCR.

The Ion AmpliSeq™ Cancer Hotspot Panel v3 will be used to detect hotspot regions of 161 oncogenes and tumor suppressor genes This research panel, with improved primer design, contains 4,648 total 4 pools (DNA pool 1: 1,891 amplicons. DNA pool 2: 1,890 amplicons. RNA pool 1: 447 amplicons. RNA pool 2: 420 amplicons.), enabling researchers to sequence challenging samples of formalin-fixed, paraffin-embedded (FFPE) tissue. Copy Number Variants (CNVs), Gene Fusions, Insertions-Deletions (indels), Single Nucleotide Polymorphisms (SNPs), Somatic Variants are identified.

HPV DNA PCR METHODOLOGY

DNA will be isolated by using QIAamp DNA mini kit (Qiagen, Hilden, Germany). The presence of HPV will be detected by using the digene® HC2 HPV DNA Test- The digene HC2 HPV DNA Test uses Hybrid Capture 2 technology to detect high-risk and low-risk HPV genotypes. It uses in vitro microplate assay based on signal-amplified nucleic acid hybridization that uses chemiluminescence for the qualitative detection of 18 types of human papillomavirus (HPV) (13 high risk and 5 low risk) DNA in cervical specimens. The test uses an RNA probe cocktail that detects 13 high-risk HPV types (16/18/31/33/35/39/45/51/52/56/58/59/68) and 5 low-risk types (6/11/42/43/44).

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven cases of primary head and neck cancers.

Exclusion Criteria:

* Patients under 18 years of age
* Pregnant and lactating women
* Multiple cancers or patients with cancer of other sites.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Histologically proven cases of Head and neck cancer undergoing treatment will be included, Next generation sequencing will be done and cohort will be followed up for 10 years
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-04-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Over all survival | 10 years
  Survival time from the diagnosis to death
Relapse free survival | 10 years
  survival time from diagnosis to recurrence or metastasis

SECONDARY OUTCOMES:
Progression free survival | 5 years
  The time from the diagnosis to progression of disease

CONTACTS AND LOCATIONS:
Overall Officials: Manoj Pandey, MS, PhD, Principal Investigator — Professor
Locations (1):
- Banaras Hindu University, Varanasi, Uttar Pradesh, India

IPD SHARING:
Plan to Share IPD: Yes
On request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 6 months
Access Criteria: On request

REFERENCES:
- [Result] Batta N, Pandey M. Mutational spectrum of tobacco associated oral squamous carcinoma and its therapeutic significance. World J Surg Oncol. 2019 Nov 27;17(1):198. doi: 10.1186/s12957-019-1741-2. PMID 31775759
- Available data/document: Mutation data — https://www.ncbi.nlm.nih.gov/clinvar/submitters/507417/ — Data of 37 mutations identified till 2020 has been uploaded, more mutations will be uploaded soon